CLINICAL TRIAL: NCT02705976
Title: Prospective Trial of a Validated Algorithm for Warfarin Dosing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Peter Brønnum, Postdoc, PhD, Aalborg University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: N-20140036
Record Dates: First submitted 2016-03-02; First posted 2016-03-11 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Anticoagulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- self-managing warfarin (Active Comparator): self-managing warfarin patients who are educated in dosing warfarin to achieve target INR value
  Interventions: Other: Active Comparator
- algorithm-suggested warfarin dosing (Experimental): algorithm-suggested warfarin dosing, where the participants are provided with a dosage suggestion of their warfarin dosage (calculated dose) to achieve target INR
  Interventions: Other: Experimental

INTERVENTIONS:
Other: Experimental — The algorithm is based on a model, which is designed to handle time series of daily warfarin intakes and INR values measured at designated time points. Based on these inputs the model is able to suggest a warfarin maintenance dose to achieve target INR value. Model parameters are initially set to population values and gradually, as data is entered into the model, these parameters become patient specific.
  Other Names: algorithm-suggested warfarin dosing
  Arms: algorithm-suggested warfarin dosing
Other: Active Comparator — Participants were (previously) educated in monitoring the INR values and to adjust the warfarin treatment accordingly to achieve a designated target INR range.
  Other Names: self-managing warfarin
  Arms: self-managing warfarin

SUMMARY:
The aim of this study is to perform a randomized trial comparing the use of the algorithm, with dosing of warfarin in standard manual dosage clinical practice, in a high quality anticoagulant setting (PSM). This is done for safety concerns and to ensure good performance of the algorithm when used in a clinical setup. The results from the study are expected to increase our knowledge of efficacy by using the algorithm in clinical practice.

ELIGIBILITY:
Inclusion Criteria

* Participants will be those ≥18 years old, must refer to Trombosecenter Aalborg and have to be educated as PSM patient
* Have to be treated for at least 1 month and willing to sign informed consent

Exclusion Criteria

* OAT treatment with phenprocoumon
* Lack of ability to handle the interface on the software used in the study (evaluated by the investigator present at the information meeting)
* Pregnancy
* Those with severe co-morbidities (e.g., creatinine > 2.5, hepatic insufficiency, active malignancy, advanced physiological age, noncompliance risk, expected survival <6 months), and physician or patient preference.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2014-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Time in therapeutic range | 6 months
  The primary study endpoint, TTR, was calculated according to the Rosendaal method

SECONDARY OUTCOMES:
Log of the variance growth rate | 6 months
  As a measure of INR variability we used log of the variance growth rate (logVGR) defined by Fihn et al.

IPD SHARING:
Plan to Share IPD: Undecided